CLINICAL TRIAL: NCT01845077
Title: Relative Bioavailability of Two Newly Developed Extended Release FDC Tablet Strengths (5mg/1000mg and 2.5 mg/750 mg) of Linagliptin/Metformin Extended Release Compared With the Free Combination of Linagliptin and Metformin Extended Release in Healthy Subjects (an Open-label, Randomised, Single Dose, Two-way Crossover Study)
Brief Title: Relative Bioavailability of 2 Fixed Dose Combinations of Linagliptin/Metformin Compared With Single Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1288.8
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin; Linagliptin

ARMS (6):
- 5 mg Linagliptin/1000 mg Metformin, fed (Active Comparator): 3 single tablets under fed conditions
  Interventions: Drug: 2x500 mg Metformin (Glumetza); Drug: 5 mg Linagliptin (Tradjenta)
- 5 mg Linagliptin/1500 mg Metformin FDC (Experimental): 2 FDC tablets under fasted conditions
  Interventions: Drug: 2 x 2.5 mg Linagliptin/750 mg Metformin FDC
- 5 mg Linagliptin/1500 mg Metformin (Active Comparator): 4 single tablets under fasted conditions
  Interventions: Drug: 3x500 mg Metformin (Glumetza); Drug: 5 mg Linagliptin (Tradjenta)
- 5 mg Linagliptin/1000 mg Metformin FDC (Experimental): 1 fixed dose combination(FDC) tablet under fasted conditions
  Interventions: Drug: 5 mg Linagliptin/1000mg Metformin FDC
- 5 mg Linagliptin/1000 mg Metformin (Active Comparator): 3 single tablets under fasted conditions
  Interventions: Drug: 5 mg Linagliptin (Tradjenta); Drug: 2 x 500 mg Metformin (Glumetza)
- 5mg Linagliptin/1000mg Metformin, FDCfed (Experimental): 1 FDC tablet under fed conditions
  Interventions: Drug: 5 mg Linagliptin/1000 mg Metformin FDC

INTERVENTIONS:
Drug: 2x500 mg Metformin (Glumetza) — 2 tablets
  Arms: 5 mg Linagliptin/1000 mg Metformin, fed
Drug: 5 mg Linagliptin/1000 mg Metformin FDC — FDC tablet
  Arms: 5mg Linagliptin/1000mg Metformin, FDCfed
Drug: 5 mg Linagliptin (Tradjenta) — 1 tablet
  Arms: 5 mg Linagliptin/1000 mg Metformin, fed
Drug: 5 mg Linagliptin (Tradjenta) — 1 tablet
  Arms: 5 mg Linagliptin/1000 mg Metformin
Drug: 3x500 mg Metformin (Glumetza) — 3 tablets
  Arms: 5 mg Linagliptin/1500 mg Metformin
Drug: 5 mg Linagliptin (Tradjenta) — 1 tablet
  Arms: 5 mg Linagliptin/1500 mg Metformin
Drug: 2 x 500 mg Metformin (Glumetza) — 2 tablets
  Arms: 5 mg Linagliptin/1000 mg Metformin
Drug: 5 mg Linagliptin/1000mg Metformin FDC — FDC Tablet
  Arms: 5 mg Linagliptin/1000 mg Metformin FDC
Drug: 2 x 2.5 mg Linagliptin/750 mg Metformin FDC — 2 FDC tablets
  Arms: 5 mg Linagliptin/1500 mg Metformin FDC

SUMMARY:
The purpose of the trial is to demonstrate the relative bioavailability of 2 newly developed fixed dose combination (FDC) tablets containing linagliptin & metformin and the single tablets of linagliptin and metformin when administered singularly.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males or females
2. Age 18 -50 years (incl)
3. Body Mass Index (BMI) 18.5 to 29.9 kg/m2 (incl.)
4. Subjects must be able to understand and comply with study requirements

Exclusion criteria:

Any deviation from healthy condition

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1288.8.1 Boehringer Ingelheim Investigational Site, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- FDC1000 Fasted, Then L+M1000 Fasted: 1 fixed dose combination (FDC) tablet 5 mg linagliptin/1000 mg metformin extended release (XR) administered on Day 1 of the first treatment period orally in the morning under fasted conditions, then 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR administered on Day 1 of the second treatment period orally in the morning under fasted conditions. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- L+M1000 Fasted, Then FDC1000 Fasted: 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR administered on Day 1 of the first treatment period orally in the morning under fasted conditions, then 1 FDC tablet 5 mg linagliptin/1000 mg metformin XR administered on Day 1 of the second treatment period orally in the morning under fasted conditions. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- FDC1000 Fed, Then L+M1000 Fed: 1 FDC tablet 5 mg linagliptin/1000 mg metformin XR administered on Day 1 of the first treatment period orally in the morning under fed conditions, then 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR administered on Day 1 of the second treatment period orally in the morning under fed conditions. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- L+M1000 Fed, Then FDC1000 Fed: 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR administered on Day 1 of the first treatment period orally in the morning under fed conditions, then 1 FDC tablet 5 mg linagliptin/1000 mg metformin XR administered on Day 1 of the second treatment period orally in the morning under fed conditions. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- FDC1500 Fasted, Then L+M1500 Fasted: 2 FDC tablets 2.5 mg linagliptin/750 mg metformin XR administered on Day 1 of the first treatment period orally in the morning under fasted conditions, then 1 tablet linagliptin 5 mg and 3 tablets metformin 500 mg XR administered on Day 1 of the second treatment period orally in the morning under fasted conditions. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- L+M1500 Fasted, Then FDC1500 Fasted: 1 tablet linagliptin 5 mg and 3 tablets metformin 500 mg XR administered on Day 1 of the first treatment period orally in the morning under fasted conditions, then 2 FDC tablets 2.5 mg linagliptin/750 mg metformin XR administered on Day 1 of the second treatment period orally in the morning under fasted conditions. Both periods lasted 4 days, separated by a washout period of at least 35 days.
Period: Treatment Period 1
Arm/Group | FDC1000 Fasted, Then L+M1000 Fasted | L+M1000 Fasted, Then FDC1000 Fasted | FDC1000 Fed, Then L+M1000 Fed | L+M1000 Fed, Then FDC1000 Fed | FDC1500 Fasted, Then L+M1500 Fasted | L+M1500 Fasted, Then FDC1500 Fasted
Started | 12 | 12 | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period
Arm/Group | FDC1000 Fasted, Then L+M1000 Fasted | L+M1000 Fasted, Then FDC1000 Fasted | FDC1000 Fed, Then L+M1000 Fed | L+M1000 Fed, Then FDC1000 Fed | FDC1500 Fasted, Then L+M1500 Fasted | L+M1500 Fasted, Then FDC1500 Fasted
Started | 12 | 12 | 12 | 12 | 12 | 12
Completed | 11 | 11 | 11 | 10 | 11 | 11
Not Completed | 1 | 1 | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0
Not completed — elevated lab values (not clinic. sign.) | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1 | 0
Period: Treatment Period 2
Arm/Group | FDC1000 Fasted, Then L+M1000 Fasted | L+M1000 Fasted, Then FDC1000 Fasted | FDC1000 Fed, Then L+M1000 Fed | L+M1000 Fed, Then FDC1000 Fed | FDC1500 Fasted, Then L+M1500 Fasted | L+M1500 Fasted, Then FDC1500 Fasted
Started | 11 | 11 | 11 | 10 | 11 | 11
Completed | 11 | 11 | 11 | 10 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) including all subjects who had been dispensed study medication and were documented to have taken at least 1 dose of study medication.
Groups:
- Total 1000 Fasted: Patients were administered 1 fixed dose combination (FDC) tablet 5 mg linagliptin/1000 mg metformin extended release (XR) orally in the morning under fasted conditions in one treatment period and 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR orally in the morning under fasted conditions in the other treatment period. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- Total 1000 Fed: Patients were administered 1 FDC tablet 5 mg linagliptin/1000 mg metformin XR orally in the morning under fed conditions in one treatment period and 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR orally in the morning under fed conditions in the other treatment period. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- Total 1500 Fasted: Patients were administered 2 FDC tablets 2.5 mg linagliptin/750 mg metformin XR orally in the morning under fasted conditions in one treatment period and 1 tablet linagliptin 5 mg and 3 tablets metformin 500 mg XR orally in the morning under fasted conditions in the other treatment period. Both periods lasted 4 days, separated by a washout period of at least 35 days.
- Total: Total of all reporting groups
Arm/Group | Total 1000 Fasted | Total 1000 Fed | Total 1500 Fasted | Total
Number analyzed (Participants) | 24 | 24 | 24 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.3) | 30.6 (9.0) | 28.4 (7.1) | 31.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 14 | 30
  Male | 16 | 16 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: AUC0-72 of Linagliptin
Description: Area Under the Concentration-time Curve of Linagliptin in Plasma Over the Time Interval 0 to 72 Hours (AUC0-72). The shown geometric coefficients of variation (gCV) are the pooled intra-individual gCV - each over 2 treatment groups (FDC1000 fasted and L+M1000 fasted, FDC1000 fed and L+M1000 fed, FDC1500 fasted and L+M1500 fasted). The geometric means are actually adjusted geometric means.
Time Frame: 1 hour (h) before drug administration and 20 minutes (min), 40 min, 1h, 1:30h, 2h, 3h, 4h, 5h, 6h, 8h, 10h, 12h, 16h, 24h, 36h, 48h and 72h after drug administration at Day 1 of each treatment period
Population: Pharmacokinetic set including all subjects of the TS who provided at least 1 observation for at least 1 primary endpoint without important protocol violations with respect to the statistical evaluation of pharmacokinetic endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- FDC1000 Fasted: 1 fixed dose combination (FDC) tablet 5 mg linagliptin/1000 mg metformin extended release (XR) administered orally in the morning of Day 1 of the corresponding treatment period under fasted conditions.
- L+M1000 Fasted: 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR administered orally in the morning of Day 1 of the corresponding treatment period under fasted conditions.
- FDC1000 Fed: 1 fixed dose combination (FDC) tablet 5 mg linagliptin/1000 mg metformin extended release (XR) administered orally in the morning of Day 1 of the corresponding treatment period under fed conditions.
- L+M1000 Fed: 1 tablet linagliptin 5 mg and 2 tablets metformin 500 mg XR administered orally in the morning of Day 1 of the corresponding treatment period under fed conditions.
- FDC1500 Fasted: 2 FDC tablets 2.5 mg linagliptin/750 mg metformin XR administered orally in the morning of Day 1 of the corresponding treatment period under fasted conditions.
- L+M1500 Fasted: 1 tablet linagliptin 5 mg and 3 tablets metformin 500 mg XR administered orally in the morning of Day 1 of the corresponding treatment period under fasted conditions
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Number analyzed (Participants) | 23 | 23 | 21 | 21 | 21 | 22
nmol*h/L | 317.0 (8.0) | 319.2 (8.0) | 309.6 (5.5) | 304.9 (5.5) | 325.8 (5.1) | 322.9 (5.1)
Statistical Analysis 1: Comparison: FDC1000 Fasted vs L+M1000 Fasted; Test type: Non-Inferiority or Equivalence — Standard acceptance criterion for bioequivalence: 90% confidence interval is completely within the bounds of 80-125%. No formal hypothesis test was conducted as study is exploratory; ANOVA; ANOVA on the logarithmic scale, adjusted for subjects within sequences as random effect and sequence, period and treatment as fixed effects; Ratio of geometric means = 99.3, 90% CI 2-sided [95.3 to 103.5]
Statistical Analysis 2: Comparison: FDC1000 Fed vs L+M1000 Fed; One patient was excluded from this analysis due to the lack of the 72h sample for the L+M1000 fed treatment; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 101.5, 90% CI 2-sided [98.4 to 104.7]
Statistical Analysis 3: Comparison: FDC1500 Fasted vs L+M1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 100.9, 90% CI 2-sided [98.2 to 103.7]

2. Primary Outcome: Cmax of Linagliptin
Description: Maximum Measured Concentration (Cmax) of Linagliptin in plasma. The shown geometric coefficients of variation (gCV) are the pooled intra-individual gCV - each over 2 treatment groups (FDC1000 fasted and L+M1000 fasted, FDC1000 fed and L+M1000 fed, FDC1500 fasted and L+M1500 fasted). The geometric means are actually adjusted geometric means.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Number analyzed (Participants) | 23 | 23 | 22 | 22 | 21 | 22
nmol/L | 10.1 (17.1) | 10.6 (17.1) | 7.7 (13.0) | 7.9 (13.0) | 11.6 (16.5) | 10.7 (16.5)
Statistical Analysis 1: Comparison: FDC1000 Fasted vs L+M1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 94.9, 90% CI 2-sided [86.8 to 103.6]
Statistical Analysis 2: Comparison: FDC1000 Fed vs L+M1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 96.8, 90% CI 2-sided [90.2 to 103.8]
Statistical Analysis 3: Comparison: FDC1500 Fasted vs L+M1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 108.6, 90% CI [99.5 to 118.5]

3. Secondary Outcome: AUC0-infinity of Linagliptin
Description: Area under the concentration-time curve of Linagliptin in plasma over the time interval from 0 extrapolated to infinity based on predicted last concentration values. The shown geometric coefficients of variation (gCV) are the pooled intra-individual gCV - each over 2 treatment groups (FDC1000 fasted and L+M1000 fasted, FDC1000 fed and L+M1000 fed, FDC1500 fasted and L+M1500 fasted). The geometric means are actually adjusted geometric means.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Number analyzed (Participants) | 23 | 23 | 22 | 22 | 21 | 22
nmol*h/L | 546.1 (12.8) | 526.5 (12.8) | 537.1 (9.6) | 510.0 (9.6) | 562.9 (13.5) | 581.1 (13.5)
Statistical Analysis 1: Comparison: FDC1000 Fasted vs L+M1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 103.7, 90% CI 2-sided [97.1 to 110.8]
Statistical Analysis 2: Comparison: FDC1000 Fed vs L+M1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 105.3, 90% CI 2-sided [99.9 to 111.0]
Statistical Analysis 3: Comparison: FDC1500 Fasted vs L+M1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 96.9, 90% CI 2-sided [90.2 to 104.1]

4. Secondary Outcome: AUC0-infinity of Metformin
Description: Area under the concentration-time curve of Metformin in plasma over the time interval from 0 extrapolated to infinity based on predicted last concentration values. The shown geometric coefficients of variation (gCV) are the pooled intra-individual gCV - each over 2 treatment groups (FDC1000 fasted and L+M1000 fasted, FDC1000 fed and L+M1000 fed, FDC1500 fasted and L+M1500 fasted). The geometric means are actually adjusted geometric means.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Number analyzed (Participants) | 23 | 23 | 22 | 23 | 21 | 22
ng*h/mL | 9037.6 (21.5) | 9326.5 (21.5) | 14031.3 (7.0) | 14069.7 (7.0) | 11037.7 (19.1) | 11512.2 (19.1)
Statistical Analysis 1: Comparison: FDC1000 Fasted vs L+M1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 96.9, 90% CI 2-sided [86.8 to 108.2]
Statistical Analysis 2: Comparison: FDC1000 Fed vs L+M1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 99.7, 90% CI 2-sided [96.1 to 103.5]
Statistical Analysis 3: Comparison: FDC1500 Fasted vs L+M1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 95.9, 90% CI 2-sided [86.7 to 106.0]

5. Primary Outcome: AUC0-tz of Metformin
Description: Area under the concentration-time curve of Metformin in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz). The shown geometric coefficients of variation (gCV) are the pooled intra-individual gCV - each over 2 treatment groups (FDC1000 fasted and L+M1000 fasted, FDC1000 fed and L+M1000 fed, FDC1500 fasted and L+M1500 fasted). The geometric means are actually adjusted geometric means.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Number analyzed (Participants) | 23 | 23 | 22 | 23 | 21 | 22
ng*h/mL | 8629.0 (21.8) | 8913.7 (21.8) | 13772.0 (7.4) | 13851.1 (7.4) | 10472.9 (18.5) | 10543.5 (18.5)
Statistical Analysis 1: Comparison: FDC1000 Fasted vs L+M1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 96.8, 90% CI 2-sided [86.6 to 108.2]
Statistical Analysis 2: Comparison: FDC1000 Fed vs L+M1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 99.4, 90% CI 2-sided [95.6 to 103.4]
Statistical Analysis 3: Comparison: FDC1500 Fasted vs L+M1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 99.3, 90% CI 2-sided [90.1 to 109.5]

6. Primary Outcome: Cmax of Metformin
Description: Maximum Measured Concentration (Cmax) of Metformin in plasma. The shown geometric coefficients of variation (gCV) are the pooled intra-individual gCV - each over 2 treatment groups (FDC1000 fasted and L+M1000 fasted, FDC1000 fed and L+M1000 fed, FDC1500 fasted and L+M1500 fasted). The geometric means are actually adjusted geometric means.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Number analyzed (Participants) | 23 | 23 | 22 | 23 | 21 | 22
ng/mL | 1047.4 (25.5) | 1085.6 (25.5) | 1119.0 (8.1) | 1084.5 (8.1) | 1347.0 (29.3) | 1250.6 (29.3)
Statistical Analysis 1: Comparison: FDC1000 Fasted vs L+M1000 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 96.5, 90% CI 2-sided [84.8 to 109.8]
Statistical Analysis 2: Comparison: FDC1000 Fed vs L+M1000 Fed; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 103.2, 90% CI 2-sided [98.9 to 107.7]
Statistical Analysis 3: Comparison: FDC1500 Fasted vs L+M1500 Fasted; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric means = 107.7, 90% CI 2-sided [92.5 to 125.4]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | FDC1000 Fasted | L+M1000 Fasted | FDC1000 Fed | L+M1000 Fed | FDC1500 Fasted | L+M1500 Fasted
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/22 | 1/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 1/23 | 1/22 | 0/23 | 3/23 | 2/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FDC1000 Fasted (N=23) | L+M1000 Fasted (N=23) | FDC1000 Fed (N=22) | L+M1000 Fed (N=23) | FDC1500 Fasted (N=23) | L+M1500 Fasted (N=23)
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FDC1000 Fasted (N=23) | L+M1000 Fasted (N=23) | FDC1000 Fed (N=22) | L+M1000 Fed (N=23) | FDC1500 Fasted (N=23) | L+M1500 Fasted (N=23)
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.